CLINICAL TRIAL: NCT05827354
Title: Incidence and Factors Associated to The Development of Post-Intensive Care Syndrome Among Family Members of Intensive Care Unit Survivors: A Longitudinal Exploratory Study
Brief Title: Incidence and Factors Associated to the Development of PICS-F Among ICU Relatives: A Longitudinal Exploratory Study
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Cristobal Padilla, Assistant Professor, School of Nursing, Pontificia Universidad Catolica de Chile
Other Study IDs: Fondecyt Iniciacion 11230203; 11230203 (Other Grant/Funding Number: ANID / FONDECYT)
Record Dates: First submitted 2023-03-29; First posted 2023-04-25 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Post Intensive Care Syndrome; Family Members; Caregiver Burden; Critical Illness; Mental Health; Physical Health; Cognitive Impairment; Family Satisfaction; Resilience; Social Support
MeSH Terms: conditions — postintensive care syndrome; Caregiver Burden; Critical Illness; Psychological Well-Being; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family Members: Family members of patients admitted to the ICU between the 1st of May 2025 and the 30th of May 2023, who survived ICU stay and are still alive up to 6 months after hospital discharge.

SUMMARY:
The constellation of long-term psychological, physical, and cognitive impairments arising after a critical illness among family members of ICU survivors has been labeled as "Post Intensive Care Syndrome - Family" (PICS-F). Despite PICS-F awareness, the long-term issues faced by ICU family members remain poorly understood with several gaps in knowledge remaining such as the role of protective psychosocial factors, caregiver burden, or family satisfaction in the development of the syndrome.

This single-center, longitudinal exploratory study, aims to determine the incidence of each PICS-F impairment (psychological, physical, and cognitive) and to identify factors (during ICU stay and after hospital discharge) associated with the development or prevention of the PICS-F impairments among family members of ICU survivors of a public hospital in Chile.

DETAILED DESCRIPTION:
During the last decades, intensive care unit (ICU) mortality rates have significantly decreased but not without adverse health-related consequences for patients and their family members. Admission to an ICU is often a stressful and traumatic experience for family members, leading to adverse psychosocial outcomes lasting beyond 12 months after hospital discharge.

The constellation of long-term psychological, physical, and cognitive impairments arising after a critical illness among family members of ICU survivors, has been labeled as "Post Intensive Care Syndrome - Family" (PICS-F). PICS-F is now being recognized as a public health burden with substantial associated costs. Despite PICS-F awareness, the long-term issues faced by ICU family members remain poorly understood with several gaps in knowledge remaining unanswered.

First, PICS-F evidence (incidence and related factors) is focused predominantly on psychological impairments with few studies exploring physical and cognitive impairments. Equally, studies on the influence of psychosocial resources (e.g., resilience, social support), which could offset PICS-F-related stress, are limited. Second, while up to 80% of the ICU family members become caregivers after the patient's hospital discharge, the effect of caregiver burden on PICS-F has received little attention. Third, is not clear the extent to which the family member´s evaluation of the ICU experience, known as family satisfaction, or other variables measured in this period can influence PICS-F.

The aim of this study is two-fold, one cross-sectional and one longitudinal aim. Among family members of ICU survivors of a public hospital in Chile, this study aims:

1. To determine the incidence of each PICS-F impairment (psychological, physical, and cognitive).
2. To identify factors associated with PICS-F impairments during ICU stay and after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

All adult family members (≥ 18 years old) identified as the patient´s representative, Spanish speakers, and likely to become responsible for providing and/or coordinating patient care after hospital discharge will be eligible.

Besides, the patient must have between 48 hours and 10 days in the ICU, be > 18 years old, and receive respiratory support (noninvasive ventilation, high-flow nasal cannula, or invasive mechanical ventilation).

Exclusion Criteria:

Family members of ICU patients with a high impending death risk (including end-of-life care / only comfort measures) or likely to be discharged from the ICU in the following 24 hours will be excluded.

Subjects (family members) will be withdrawn from the study at any point if the patient dies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Family members of ICU survivors in a public hospital in Santiago, Chile who meet the inclusion criteria will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of psychological impairment in family members of ICU survivors | 3 months after hospital discharge
  Symptoms of anxiety and depression (1) or Post-traumatic stress disorder (PTSD) (2) (1 or 2):
  1. Anxiety and depressive symptoms measured using the 4-item version of the Patient Health Questionnaire (PHQ - 4), summed score range from 0 (best) to 12 (worst). Presence of symptoms of anxiety and depression if summed PHQ - 4 score ≥ 6.
  2. PTSD symptoms measured using the 6-item version of the Impact of Event Scale (IES - 6), summed score range from 0 (best) to 24 (worst). Presence of PTSD symptoms if averaged IES - 6 score ≥ 1.75.
Incidence of psychological impairment in family members of ICU survivors | 6 months after hospital discharge
  Symptoms of anxiety and depression (1) or Post-traumatic stress disorder (PTSD) (2) (1 or 2):
  1. Anxiety and depressive symptoms measured using the 4-item version of the Patient Health Questionnaire (PHQ - 4), summed score range from 0 (best) to 12 (worst). Presence of symptoms of anxiety and depression if summed PHQ - 4 score ≥ 6.
  2. PTSD symptoms measured using the 6-item version of the Impact of Event Scale (IES - 6), summed score range from 0 (best) to 24 (worst). Presence of PTSD symptoms if averaged IES - 6 score ≥ 1.75.
Incidence of physical impairment in family members of ICU survivors | 3 months after hospital discharge
  Symptoms of clinically significant fatigue. Clinical fatigue measured using 4 items of the "energy/fatigue" subscale (Vt) of the Short Form Health Survey (SF - 36). Averaged score range from 100 (best) to 0 (worst): Presence of clinical fatigue if averaged SF - 36 Vt score < 45.
Incidence of physical impairment in family members of ICU survivors | 6 months after hospital discharge
  Symptoms of clinically significant fatigue. Clinical fatigue measured using 4 items of the "energy/fatigue" subscale (Vt) of the Short Form Health Survey (SF - 36). Averaged score range from 100 (best) to 0 (worst): Presence of clinical fatigue if averaged SF - 36 Vt score < 45.
Incidence of cognitive impairment in family members of ICU survivors | 3 months after hospital discharge
  Cognitive impairment measured using the memory, fluency, and orientation (MEFO) test. Summed score range from 13 (best) to 0 (worst). Presence of cognitive impairment if summed MEFO test score < 9.
Incidence of cognitive impairment in family members of ICU survivors | 6 months after hospital discharge
  Cognitive impairment measured using the memory, fluency, and orientation (MEFO) test. Summed score range from 13 (best) to 0 (worst). Presence of cognitive impairment if summed MEFO test score < 9.

SECONDARY OUTCOMES:
Symptoms of Anxiety and Depression in family members of ICU survivors | Between the 3rd - 7th day of ICU admission
  Anxiety and depressive symptoms measured using the PHQ - 4, summed score range, 0 (best) to 12 (worst)): Presence of symptoms of anxiety and depression if summed PHQ - 4 score ≥ 6.
Symptoms of Anxiety and Depression in family members of ICU survivors | Up to 1 week after ICU discharge
  Anxiety and depressive symptoms measured using the PHQ - 4, summed score range, 0 (best) to 12 (worst)): Presence of symptoms of anxiety and depression if summed PHQ - 4 score ≥ 6.
Symptoms of PTSD in family members of ICU survivors | Up to 1 week after ICU discharge
  PTSD-related symptoms measured using the IES - 6, summed score range from 0 (best) to 24 (worst)): Presence of PTSD symptoms if averaged IES - 6 score ≥ 1.75.
Physical impairment in family members of ICU survivors | Between the 3rd - 7th day of ICU admission
  Symptoms of clinically significant fatigue. Clinical fatigue measured using 4 items of the "energy/fatigue" subscale (Vt) of SF - 36. Averaged score range from 100 (best) to 0 (worst): Presence of clinical fatigue if averaged SF - 36 Vt score < 45.
Physical impairment in family members of ICU survivors | Up to 1 week after ICU discharge
  Symptoms of clinically significant fatigue. Clinical fatigue measured using 4 items of the "energy/fatigue" subscale (Vt) of SF - 36. Averaged score range from 100 (best) to 0 (worst): Presence of clinical fatigue if averaged SF - 36 Vt score < 45.
Cognitive impairment in family members of ICU survivors | Between the 3rd - 7th day of ICU admission
  Cognitive impairment measured using the MEFO test. Summed score range from 13 (best) to 0 (worst). Presence of cognitive impairment if summed MEFO test score < 9.
Cognitive impairment in family members of ICU survivors | Up to 1 week after ICU discharge
  Cognitive impairment measured using the MEFO test. Summed score range from 13 (best) to 0 (worst). Presence of cognitive impairment if summed MEFO test score < 9.
Perceived Social Support in family members of ICU survivors | Between the 3rd - 7th day of ICU admission
  Perceived social support measured using the modified 8-item version of the Medical Outcomes Study Social Support Survey (mMOS - SSS). Averaged score range from 100 (best) to 0 (worst).
Perceived Social Support in family members of ICU survivors | Up to 1 week after ICU discharge
  Perceived social support measured using the modified 8-item version of the Medical Outcomes Study Social Support Survey (mMOS - SSS). Averaged score range from 100 (best) to 0 (worst).
Perceived Social Support in family members of ICU survivors | 3 months after hospital discharge
  Perceived social support measured using the modified 8-item version of the Medical Outcomes Study Social Support Survey (mMOS - SSS). Averaged score range from 100 (best) to 0 (worst).
Perceived Social Support in family members of ICU survivors | 6 months after hospital discharge
  Perceived social support measured using the modified 8-item version of the Medical Outcomes Study Social Support Survey (mMOS - SSS). Averaged score range from 100 (best) to 0 (worst).
Resilience in family members of ICU survivors | Between the 3rd - 7th day of ICU admission
  Resilience measured using the Brief Resilient Coping Scale (BRCS). Summed score range from 20 (best) to 4 (worst). Presence of low resilience if summed BRCS score ≤ 13.
Resilience in family members of ICU survivors | Up to 1 week after ICU discharge
  Resilience measured using the Brief Resilient Coping Scale (BRCS). Summed score range from 20 (best) to 4 (worst). Presence of low resilience if summed BRCS score ≤ 13.
Resilience in family members of ICU survivors | 3 months after hospital discharge
  Resilience measured using the Brief Resilient Coping Scale (BRCS). Summed score range from 20 (best) to 4 (worst). Presence of low resilience if summed BRCS score ≤ 13.
Resilience in family members of ICU survivors | 6 months after hospital discharge
  Resilience measured using the Brief Resilient Coping Scale (BRCS). Summed score range from 20 (best) to 4 (worst). Presence of low resilience if summed BRCS score ≤ 13.
Family Satisfaction in family members of ICU survivors | Between the 3rd - 7th day of ICU admission
  Family satisfaction measured using the Family Satisfaction with Care in the Intensive Care Unit - 24 (FS ICU - 24). Averaged score range from 100 (best) to 0 (worst).
Family Satisfaction in family members of ICU survivors | Up to 1 week after ICU discharge
  Family satisfaction measured using the Family Satisfaction with Care in the Intensive Care Unit - 24 (FS ICU - 24). Averaged score range from 100 (best) to 0 (worst).
Caregiver Burden in family members of ICU survivors | 3 months after hospital discharge
  Caregiver Burden measured using the 7-item version of the ZARIT Burden Interview (ZBI). Summed score range from 7 (best) to 35 (worst). Presence of intense caregiver burden if summed ZBI score ≥ 17.
Caregiver Burden in family members of ICU survivors | 6 months after hospital discharge
  Caregiver Burden measured using the 7-item version of the ZARIT Burden Interview (ZBI). Summed score range from 7 (best) to 35 (worst). Presence of intense caregiver burden if summed ZBI score ≥ 17.
Functional Independence in ICU survivors | Between the 3rd - 7th day of ICU admission (prior ICU admission status)
  Patient´s functional independence using the Barthel Index (BI). Summed score range from 100 (best) to 0 (worst)
Functional Independence in ICU survivors | Up to 1 week after ICU discharge
  Patient´s functional independence using the Barthel Index (BI). Summed score range from 100 (best) to 0 (worst)
Functional Independence in ICU survivors | 3 months after hospital discharge
  Patient´s functional independence using the Barthel Index (BI). Summed score range from 100 (best) to 0 (worst)
Functional Independence in ICU survivors | 6 months after hospital discharge
  Patient´s functional independence using the Barthel Index (BI). Summed score range from 100 (best) to 0 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Padilla F., PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Dra. Eloisa I. Diaz, La Florida, RM, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Beusekom I, Bakhshi-Raiez F, de Keizer NF, Dongelmans DA, van der Schaaf M. Reported burden on informal caregivers of ICU survivors: a literature review. Crit Care. 2016 Jan 21;20:16. doi: 10.1186/s13054-016-1185-9. PMID 26792081
- [Background] Rawal G, Yadav S, Kumar R. Post-intensive Care Syndrome: an Overview. J Transl Int Med. 2017 Jun 30;5(2):90-92. doi: 10.1515/jtim-2016-0016. eCollection 2017 Jun. PMID 28721340
- [Background] Kean S, Smith GD. Editorial: surviving critical illness: intensive care and beyond. J Clin Nurs. 2014 Mar;23(5-6):603-4. doi: 10.1111/jocn.12555. No abstract available. PMID 24589228
- [Background] Davidson JE, Harvey MA. Patient and Family Post-Intensive Care Syndrome. AACN Adv Crit Care. 2016 Apr-Jun;27(2):184-6. doi: 10.4037/aacnacc2016132. No abstract available. PMID 27153307
- [Background] Johnson CC, Suchyta MR, Darowski ES, Collar EM, Kiehl AL, Van J, Jackson JC, Hopkins RO. Psychological Sequelae in Family Caregivers of Critically III Intensive Care Unit Patients. A Systematic Review. Ann Am Thorac Soc. 2019 Jul;16(7):894-909. doi: 10.1513/AnnalsATS.201808-540SR. PMID 30950647
- [Background] Choi J, Tate JA, Hoffman LA, Schulz R, Ren D, Donahoe MP, Given BA, Sherwood PR. Fatigue in family caregivers of adult intensive care unit survivors. J Pain Symptom Manage. 2014 Sep;48(3):353-63. doi: 10.1016/j.jpainsymman.2013.09.018. Epub 2014 Jan 16. PMID 24439845
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] Cameron JI, Chu LM, Matte A, Tomlinson G, Chan L, Thomas C, Friedrich JO, Mehta S, Lamontagne F, Levasseur M, Ferguson ND, Adhikari NK, Rudkowski JC, Meggison H, Skrobik Y, Flannery J, Bayley M, Batt J, dos Santos C, Abbey SE, Tan A, Lo V, Mathur S, Parotto M, Morris D, Flockhart L, Fan E, Lee CM, Wilcox ME, Ayas N, Choong K, Fowler R, Scales DC, Sinuff T, Cuthbertson BH, Rose L, Robles P, Burns S, Cypel M, Singer L, Chaparro C, Chow CW, Keshavjee S, Brochard L, Hebert P, Slutsky AS, Marshall JC, Cook D, Herridge MS; RECOVER Program Investigators (Phase 1: towards RECOVER); Canadian Critical Care Trials Group. One-Year Outcomes in Caregivers of Critically Ill Patients. N Engl J Med. 2016 May 12;374(19):1831-41. doi: 10.1056/NEJMoa1511160. PMID 27168433
- [Background] Nadig N, Huff NG, Cox CE, Ford DW. Coping as a Multifaceted Construct: Associations With Psychological Outcomes Among Family Members of Mechanical Ventilation Survivors. Crit Care Med. 2016 Sep;44(9):1710-7. doi: 10.1097/CCM.0000000000001761. PMID 27065467
- [Background] Haines KJ, Denehy L, Skinner EH, Warrillow S, Berney S. Psychosocial outcomes in informal caregivers of the critically ill: a systematic review. Crit Care Med. 2015 May;43(5):1112-20. doi: 10.1097/CCM.0000000000000865. PMID 25654174
- [Background] Padilla Fortunatti C, De Santis JP, Munro CL. Family Satisfaction in the Adult Intensive Care Unit: A Concept Analysis. ANS Adv Nurs Sci. 2021 Oct-Dec 01;44(4):291-305. doi: 10.1097/ANS.0000000000000360. PMID 33624988
- [Background] Beesley SJ, Hirshberg EL, Wilson EL, Butler JM, Oniki TA, Kuttler KG, Orme JF, Hopkins RO, Brown SM. Depression and Change in Caregiver Burden Among Family Members of Intensive Care Unit Survivors. Am J Crit Care. 2020 Sep 1;29(5):350-357. doi: 10.4037/ajcc2020181. PMID 32869070
- [Derived] Padilla-Fortunatti C, Rojas-Silva N, Cortes-Maripangue S, Palmeiro-Silva Y, Rojas-Jara V, Nilo-Gonzalez V, Cifuentes-Avendano B, Morales-Morales D, Garces-Brito N. Incidence and factors associated with post-intensive care syndrome among caregivers of intensive care unit survivors: Protocol for a cohort study. PLoS One. 2025 May 16;20(5):e0324013. doi: 10.1371/journal.pone.0324013. eCollection 2025. PMID 40378139